CLINICAL TRIAL: NCT02771769
Title: A Multi-center Prospective Study to Analyze Cancer-derived Cell-free DNA (cfDNA) in Men With Elevated PSA Levels
Brief Title: Analysis of Cell-free DNA (cfDNA) in Men With Elevated PSA Levels
Status: Terminated | Type: Observational
Why Stopped: Data review
Sponsor: Chronix Biomedical Corporation (Industry)
Collaborators: Smerud Medical Research International AS (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: CHX-2015-01
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Prostatic Neoplasms
Keywords: cell-free DNA; copy number instability; liquid biopsy; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell-free and cell-associated DNA will be obtained from plasma and peripheral blood mononuclear cells, respectively. DNA will be stored until study is completed and data are published.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood draw — Participants will have a venous blood draw of ~20mLs before prostate biopsy. The biopsy will then be performed and histologically graded for any malignancy present. This grade will be statistically analyzed with respect to the Copy Number Instability (CNI) determined from the results of the molecular examination of the cell-free DNA in the blood.

SUMMARY:
This is a multi-centre prospective study in which blood samples will be taken from 1500 male patients aged between 21-80 scheduled for prostate biopsy. Analysis of cell-free cancer DNA extracted from these samples will be undertaken to determine whether copy number instability scores derived from the cfDNA correlates with PSA screening levels and prostate biopsy results (i.e. Gleason score) in these patients.

DETAILED DESCRIPTION:
The prostate is the most common site of cancer in men with 240,000 new cases diagnosed annually in the United States with approximately 28,000 yearly deaths. Prostate screening typically relies on digital rectal exam (DRE) and prostate specific antigen (PSA) levels. Limitations of the PSA test include its low sensitivity and low specificity and its inability to distinguish between low-grade and high-grade lesions. Recent screening trials suggest that PSA-based screening programs result in small or no reduction in mortality, and have significant treatment-related adverse events (AEs). Better serum/plasma biomarkers are needed to supplement the PSA test in the diagnosis and management of a disease with a multiplicity of presentations and clinical outcomes.

Cancer-derived DNA present in peripheral blood (referred to as cell-free DNA or cfDNA) was first reported in 1948, but research into this area remained in a dormant state for over 50 years. Over the last ten years however, the development of Next Generation Sequencing (NGS) using massive parallel arrays has allowed researchers to create a database robust enough to distinguish normal genomic from non-diploid cfDNA. In 2008, fetal trisomy of chromosome 21 was detected by analyzing cfDNA in maternal blood. Since then, the method has been validated for trisomy 13, 18, and 21 as a clinical laboratory procedure with remarkable accuracy >99%. Recently, cancer derived cfDNA has been demonstrated to recapitulate genomic tumor DNA. Current clinical acceptance of the utility of cfDNA in cancer diagnosis has been demonstrated in multiple abstracts at the 2014 and 2015 ASCO meetings in Chicago.

In a recent publication in Clinical Chemistry, researchers at Vanderbilt University, Gottingen, Germany, and at the University of Toronto, Canada, analyzed cfDNA in the bloodstream from healthy controls as compared to those with clinically diagnosed prostate cancer. The results of this study demonstrated that it is possible to distinguish prostate cancer from healthy controls without prior knowledge of the genetic signature of the tumors and with over three times the sensitivity of the FDA-approved blood test for prostate cancer (i.e., prostate-specific antigen (PSA)). The study examined serum from more than 200 subjects with prostate cancer and more than 200 controls. The comparative data included PSA levels and prostate tissue biopsy grading (referred to as the Gleason score). The technique distinguished prostate cancer from normal controls with 84% accuracy and cancer from benign hyperplasia and prostatitis with an accuracy of 91%. Because the method quantifies the inherent chromosomal instability of cancer and can be followed as a function of time (without having to do an invasive tissue biopsy), it is called a "liquid biopsy." This multi-centre clinical study will analyze cfDNA from subjects scheduled for prostate biopsy and is designed to validate the results obtained in the above-mentioned retrospective study. If validated, the prostate cfDNA determination test will provide a non-invasive test to aid in the diagnosis of prostate cancer, as well as provide guidance on whether a biopsy should be performed.

With regard to the study procedures used, the study subject will undergo routine venipuncture and ~20 millilitres of blood (approximately 2 tablespoons) will be collected. The blood will then be processed by the Sponsor's laboratory and sent to the Sponsor's testing facility in Gottingen, Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Who, in the opinion of the site Investigator, have an abnormal PSA level as measured by a CLIA certified laboratory or non-USA equivalent within the last 60 days, and/or
2. Who, in the opinion of the site Investigator, have an abnormal digital rectal examination

Exclusion Criteria:

1. Male subjects with active or historical histologically confirmed diagnosis of malignancy
2. Male subjects who have participated in a clinical trial involving an investigational drug within the 28 days prior to signing the informed consent form

Ages: 21 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male subjects between the ages of 21-80 who are scheduled for a prostate biopsy and meet one of the eligibility criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01; Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
CNI correlation with biopsy | Through completion of study and all data analysis which may take up to 2 years.
  To determine if copy number instability (CNI scores) derived from analysis of cell-free cancer DNA (cfDNA) in patients undergoing prostate biopsy correlates with biopsy diagnosis of prostate cancer.

SECONDARY OUTCOMES:
CNI correlation with BPH | Through completion of study and all data analysis which may take up to 2 years.
  To determine if copy number instability (CNI scores) derived from analysis of cell-free DNA (cfDNA) in patients undergoing prostate biopsy can distinguish between biopsy diagnosis of benign prostatic hyperplasia (BPH) and prostate cancer.
CNI correlation with PIN | Through completion of study and all data analysis which may take up to 2 years.
  To determine if copy number instability (CNI scores) derived from analysis of cell-free DNA (cfDNA) in patients undergoing prostate biopsy correlates with measured evidence of prostatic intraepithelial neoplasia (PIN).

CONTACTS AND LOCATIONS:
Overall Officials: David F Penson, MD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - University of Maryland Cancer Center, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Participants may request data upon writing to their physician. Data will not be available until after publication of data.

REFERENCES:
- [Result] Chou R, Croswell JM, Dana T, Bougatsos C, Blazina I, Fu R, Gleitsmann K, Koenig HC, Lam C, Maltz A, Rugge JB, Lin K. Screening for prostate cancer: a review of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2011 Dec 6;155(11):762-71. doi: 10.7326/0003-4819-155-11-201112060-00375. Epub 2011 Oct 7. PMID 21984740
- [Result] Bill-Axelson A, Holmberg L, Garmo H, Rider JR, Taari K, Busch C, Nordling S, Haggman M, Andersson SO, Spangberg A, Andren O, Palmgren J, Steineck G, Adami HO, Johansson JE. Radical prostatectomy or watchful waiting in early prostate cancer. N Engl J Med. 2014 Mar 6;370(10):932-42. doi: 10.1056/NEJMoa1311593. PMID 24597866
- [Result] Renard E, Bringer J, Augustin I, Orsetti A, Jaffiol C. [Value of dexamethasone suppression tests in the diagnosis of hypercortisolism of ectopic or adrenal origin]. Presse Med. 1989 Feb 25;18(8):435. No abstract available. French. PMID 2540489